CLINICAL TRIAL: NCT06129916
Title: Assessing the Acceptability, Feasibility, Effectiveness and Cost-effectiveness of Long-acting Depot Buprenorphine (LADB) for the Treatment of Opioid Dependence in Low- and Middle-income Countries (LMIC): a Multicentre International Study
Brief Title: Assessing the Acceptability, Feasibility, Effectiveness and Cost-effectiveness of LADB
Status: Not yet recruiting | Type: Observational
Sponsor: PATH (Other)
Collaborators: UNITAID (Other); World Health Organization (Other); Médecins du Monde (Other); Frontline AIDS (Other); London School of Hygiene and Tropical Medicine (Other); International Network of People who Use Drugs (Unknown); Monash University (Other); Population Services International (Other); Burnet Institute (Other); University of Bristol (Other); Alliance for the Public's Health (Other); Coact Technical Support Limited (Unknown)
Responsible Party: Sponsor
Other Study IDs: RES-00617
Record Dates: First submitted 2023-10-04; First posted 2023-11-13 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PWID who opt for LADB: People with opioid dependence who opt to initiate LADB across a range of LMIC settings over a 48-week period
  Interventions: Drug: long-acting depot buprenorphine (LADB)
- PWID who opt for standard of care: People with opioid dependence who refuse to initiate LADB and opt for standard of care

INTERVENTIONS:
Drug: long-acting depot buprenorphine (LADB) — The intervention will measure patient-centered outcomes in people initiating LADB among a cohort of opioid-dependent PWID across sites in the seven project LMIC. Study participants will be enrolled from selected clinics that deliver routine opioid agonist maintenance treatment to PWID. The intervention will 1) Compare characteristics at baseline of those service clients who do and do not initiate LADB in relation to demographic characteristics, history of drug use, and outcomes; 2) Measure side effects and adverse events among those initiating LADB; and 3) Where appropriate, assess changes in outcomes between time of LADB initiation and 48 week follow-up, including HCV and HIV testing and treatment, quality of life, employment opportunities, and service preferences.
  Groups: PWID who opt for LADB

SUMMARY:
The goal of the proposed study is to generate evidence on the acceptability, feasibility, effectiveness, and cost-effectiveness of introducing long-acting depot buprenorphine (LADB) as an additional option for the treatment of opioid dependence in low- and middle-income countries (LMIC) among people who inject drugs (PWID) with opioid dependence. The study results will be used to inform global and local policies and guidelines to introduce LADB as a treatment option and to advocate for access to a sustainable supply of LADB in LMIC.

DETAILED DESCRIPTION:
Despite the proven effectiveness of opioid agonist maintenance treatment (OAMT), its coverage and use remain low globally and, particularly, in low- and middle-income countries (LMIC), in part due to challenges related to limited choice of OAMT medication and dosing options. The long-acting depot buprenorphine (LADB) formulation of OAMT, with either weekly or monthly administration, could provide a more discreet, convenient, and less stigmatizing form of treatment and the potential to improve client retention in care, as well as economic stability. It therefore may address unmet need among individuals who could benefit from OAMT and are not already taking it or who would prefer a long-acting option over current OAMT options. Studies have demonstrated the effectiveness and acceptability of LADB among those with opioid dependence in high-income settings. However, there are no known such studies conducted in LMIC.

The aim of the study is to determine the acceptability, feasibility, effectiveness, public health impact, and cost-effectiveness of introducing LADB in a range of LMIC.

The study will collect data from participants with opioid use disorder, service providers, and health policymakers/decision-makers across seven diverse LMIC: Egypt, India, Kyrgyzstan, South Africa, Tanzania, Ukraine, and Vietnam.

This is a multicenter, mixed-method study designed with community engagement and co-production. The study consists of four interlinked modules: Module 1 (feasibility) includes a process evaluation to monitor implementation and assess barriers, drawing on program data and interviews with service providers and other key stakeholders; Module 2 (effectiveness) involves a prospective cohort choice study among people with opioid dependence, initiating LADB and following up over 48 weeks; Module 3 (values and preferences, plus acceptability) includes key informant interviews and focus group discussions with people with opioid dependence to understand overall acceptability, values, preferences, experiences, and concerns relating to LADB; Module 4 (public health impact and cost-effectiveness) involves modeling based on collected data to estimate impact and cost-effectiveness of LADB in LMIC settings.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years old or older.
* Are verified (by certified clinician) opioid dependents according to the International Classification of Diseases 11th Revision.
* Are not pregnant (verified by screening).
* Are eligible to receive OAMT at a participating site.
* Consent to attend the clinic and adhere to clinical protocols
* Have the capacity to consent to participating in research.
* Provide written informed consent.

Exclusion Criteria:

* Have a history or presence of an allergic or adverse response (including rash or anaphylaxis) to BUP or the Atrigel® delivery system (a registered trademark of Tolmar Therapeutics Inc.) if Sublocade is chosen.
* Have any contraindication to BUP or methadone.
* Show signs of clinically significant medical conditions which would compromise compliance with the protocol and/or client safety in line with clinical guidelines for the administration of injectable BUP for OAMT.
* Are currently taking oral or depot naltrexone therapy or are enrolled in any form of naltrexone therapy within 30 or 90 days prior to study screening, respectively.
* Are in thepost partum period (defined as 6 weeks) or confirmed as pregnant.
* Have an inability or unwillingness to provide informed consent or abide by the requirements of the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Sites will set a target for participation among women in line with the percentage of women accessing needle/syringe programmes and OAMT locally. Where data are not currently available on gender or if attendance is very low, we aim to recruit a minimum quota of 10% to ensure meaningful participation among women.
Study Population: The study will collect data from participants with opioid use disorder across eight diverse LMIC: Egypt, India, Kyrgyzstan, Nigeria, South Africa, Tanzania, Ukraine, and Vietnam.
Sampling Method: Non-Probability Sample
Enrollment: 760 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment Satisfaction Questionnaire for Medication 1.4 assessed through patient reported outcomes on effectiveness, side-effects, convenience and global satisfaction in relation to the medication | 48 weeks
  The primary measure for treatment satisfaction will be collected through the Treatment Satisfaction Questionnaire for Medication 1.4 at 48 weeks. This is a generic measure of treatment satisfaction with medication. It has 14 questions divided into subscales (effectiveness; side effects, convenience and global satisfaction). Response are on a Likert-scale of 5 or 7 points except for 1 yes/no question on the presence of side effects. The scores are calculated for each of the subscales, which range from 0 to100 with higher scores indicating higher patient satisfaction with medication.
Retention in Care | 48 weeks
  The primary measure for retention in care will be estimated as the proportion of people on LADB at 48 weeks
Nonmedical opioid use | 48 weeks
  Assess degree of non-medical opioid use in the last month measured at week 48, in terms of number of days that non-medical opioids were not used in the last 4 weeks.

SECONDARY OUTCOMES:
% of participants who have received testing for HIV and Hepatitis C (HCV) at 48 weeks, frequency of testing, % testing positive for antibodies to HIV or HCV and % linked to treatment and % retained into treatment | 48 weeks
  Retention into HIV treatment will be measured through self-report using a predefined threshold of adherence (80 to 100%) in consultation with sites as well as through recoding return visits for medication refills. Retention into HCV treatment will be measured as the proportion of those completing treatment and who have sustained virologic response 12 weeks after treatment. These data will be extracted from clinical records at programme sites.
% of participants with self reported symptoms of depression at 48 weeks. | 48 weeks
  Measured through the self-completion scale (PHQ-9 [9-question Patient Health Questionnaire] with scale from 0-3, lower score indicating better mental health
% of participants with self-reported symptoms of anxiety at 48 weeks. | 48 weeks
  Measured through the self-completion scale GAD-7 [Generalized Anxiety Disorder 7) with scale from 0-3, lower score indicating better mental health
% of participants reporting recent thoughts of or attempts at suicide at 48 weeks. | 48 weeks
  This will be taken from other studies among people who inject drugs with "suicidality" specified as recent (within last 4 weeks) thoughts of and attempts at suicide.
Patient-reported outcomes using the EuroQol measures of health status | 48 weeks
  Patient-reported outcomes (PROMs) assessing health-related quality of life will include the EQ5D-5L, which measures the five dimensions of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression (range 1-5, lower score indicates better health)
Patient-reported outcomes using the EuroQol visual analogue scale (EQVAS) | 48 weeks
  Patient-reported outcomes (PROMs) assessing health-related quality of life using a visual analogue scale EQVAS (range 0-100, higher score indicates better health).
% of participants reporting a non-fatal overdose in the last 6 months | 48 weeks
  This will be defined as losing consciousness due to a drug-related overdose (opioids or ATS) in the last 6 months.
% of participants reporting risky levels of alcohol use (range 0-12, higher score indicates higher risk alcohol use). | 48 weeks
  Self-reported alcohol use will be measured using the Alcohol Use Disorders Identification Test (AUDIT)
% of participants reporting experience of Stigma and discrimination is measured through the substance use stigma mechanism scale (SU-SMS) (range 1-5, higher scores denote greater stigma and discrimination) | 48 weeks
  Stigma and discrimination will be measured using the substance use stigma mechanism scale that measures enacted and internalized stigma from family and health care workers.
% of participants reporting being arrested by the police in the last 6 months measured at 48 weeks. | 48 weeks
  This is a self reported measure: "In the last 6 months, have you been arrested or detained or charged by police in (XX location) for any reason?"
% of participants who have been in prison in the last 6 months measured at 48 weeks | 48 weeks
  This is a self-reported measure: "In the last 6 months, have you spent time in prison, jail or a young offenders institute?"

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Green, Principal Investigator — PATH

IPD SHARING:
Plan to Share IPD: No